CLINICAL TRIAL: NCT02951546
Title: Body Composition, Adiposity Phenotype, Metabolic Flexibility, and Gut Microbiota in PNPLA3 and TM6SF2 Gene Variant Carriers and Non-carriers With Nonalcoholic Fatty Liver Disease. Effects of a Nutritional Intervention Combined to Exercise
Brief Title: Metabolic Flexibility, Gut Microbiota, Healthy Diet and Exercise in NAFLD on Genetics Base
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other); Università degli studi di Roma Foro Italico (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, STEFANO GINANNI CORRADINI, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RIF.CE:4119
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet, Mediterranean; Diet, Fat-Restricted; Exercise

STUDY DESIGN:
Intervention Model Description: Nonalcoholic fatty liver disease (NAFLD) is associated to obesity, metabolic syndrome and genetic predisposition: specific variants of the genes PNPLA3 and TM6SF2 are the most involved. Also biochemical mechanisms that affect the "metabolic flexibility" need to be better clarified.
  It is known that a dietary intervention and a physical personalized training, reduce either the hepatic fat content either insulin resistance.
  Therefore, the aim of the study is to evaluate "metabolic flexibility" in obese NAFLD subjects taking in account the presence or absence of PNPLA3 and TM6SF2 polymorphism and the histopathological diagnosis of either simple steatosis or nonalcoholic steatohepatitis (NASH). The composition of gut microbiota will be also evaluated.
  Finally, two distinct healthy dietary profiles accompanied by a personalized physical training, will be tested to comprehend whether and how "healthy diets" could operate in the clinical treatment of NAFLD and related conditions.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mediterranean diet (Experimental): Hypocaloric Mediterranean diet for a 4-month period;
  Aerobic exercise training for a 4-month period;
  Interventions: Dietary Supplement: Mediterranean diet; Other: Aerobic exercise
- Low fat diet (Experimental): Hypocaloric low fat diet supplemented by branched and essential amino acids considering the total protein intake for a 4- month period;
  Aerobic exercise training for a 4- month period;
  Interventions: Dietary Supplement: Low fat diet; Other: Aerobic exercise

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — In the Mediterranean diet fat intake will be equal to 35% of the total energy intake minus carbohydrate and protein energy carbohydrate as 65% of total calorie intake, dietary cholesterol <300 mg/day, dietary fiber 25 g/day.
  Arms: Mediterranean diet
Dietary Supplement: Low fat diet — In the hypocaloric low fat diet, fat will represent less than 25% of the total energy intake. Branched and essential amino acids will be administered taking into account the total protein intake.
  Arms: Low fat diet
Other: Aerobic exercise — A personalized program of aerobic exercise will be prescribed to the participants of both arms, following the "FITT" principles (frequency, intensity, time and type).

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is associated to obesity, metabolic syndrome and genetic predisposition: specific variants of the genes PNPLA3 and TM6SF2 are the most involved. Also biochemical mechanisms that affect the "metabolic flexibility" need to be better clarified.

It is known that a dietary intervention, accompanied by a physical personalized training, reduce either the hepatic fat content either insulin resistance.

Therefore, the aim of the study is to evaluate "metabolic flexibility" in obese NAFLD subjects taking in account the presence or absence of PNPLA3 and TM6SF2 polymorphism and the histopathological diagnosis of either simple steatosis or nonalcoholic steatohepatitis (NASH). The composition of gut microbiota will be also evaluated.

Finally, two distinct healthy dietary profiles accompanied by a personalized physical training, will be tested to comprehend whether and how "healthy diets" could operate in the clinical treatment of NAFLD and related conditions.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is frequently associated to obesity and metabolic syndrome. In NAFLD, a heritable component to disease susceptibility has been demonstrated: the variants of the genes PNPLA3 and TM6SF2 are the most involved genetic determinants.

To date, biochemical mechanisms that affect the "metabolic flexibility" in obese NAFLD subjects, in presence or absence of genetic susceptibility, need to be better clarified.

Different studies demonstrated that a dietary intervention, accompanied by a physical personalized training, significantly reduce either the hepatic fat content either insulin resistance in overweight and obese subjects, independently of weight loss.

On these bases, the aim of the study is to evaluate "metabolic flexibility" in obese NAFLD subjects taking in account their genetics (presence or absence of PNPLA3 and TM6SF2 polymorphisms) and the histopathological diagnosis of either simple steatosis or nonalcoholic steatohepatitis (NASH). In addition, the composition of gut microbiota will be evaluated.

Finally, in this study, two distinct healthy dietary profiles accompanied by a personalized physical training, will be tested in order to comprehend whether and how "healthy diets" could be effective not only in the prevention, but also in the clinical treatment of NAFLD and other related conditions.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) > 30 Kg/m2 and < 40 Kg/m2;
* Caucasian Italian subjects
* hepatic steatosis according with ultrasonographic Hamaguchi's criteria and/or hypertransaminasemia (ALT >30 IU/L in men and >20 IU/L in women)

Exclusion Criteria:

* any malignant disease during the last 5 years;
* any inflammatory or autoimmune disease;
* corticosteroids for systemic use;
* renal failure (GFR<90 ml/min);
* heart failure (NYHA classes II-IV);
* history of viral or autoimmune liver disease;
* any cause cirrhosis;
* excessive alcohol intake (>140g/week for men and 70g/week for women);
* participation in a reducing-weight program in the last 3 months;
* level of physical activity higher than 3 METs;
* therapy with antibiotics during the last 3 months;
* bile salts, cholestyramine during the last 6 months before enrollment;
* previous cholecystectomy;
* gallbladder disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Cholesterol assessment | baseline
  total cholesterol, HDL- cholesterol, LDL- cholesterol levels reported as mg/dl
Cholesterol assessment | 18 weeks after baseline
  total cholesterol, HDL- cholesterol, LDL- cholesterol levels reported as mg/dl
triglycerides assessment | baseline
  tryglicerides levels reported as mg/dl
triglycerides assessment | 18 weeks after baseline
  tryglicerides levels reported as mg/dl
metabolic flexibility variation in liver function; | baseline
  alanine aminotransferase (ALT) [U/L] , aspartate aminotransferase (AST) [UI/L]
metabolic flexibility variation in liver function; | 18 weeks after baseline
  alanine aminotransferase (ALT) [U/L] , aspartate aminotransferase (AST) [UI/L]
Waist circumference measurements; | baseline
  waist circumference reported as cm
Waist circumference measurements; | 18 weeks after baseline
  waist circumference reported as cm
anthropometric measurements; | baseline
  Body mass index reported as kg/m^2
anthropometric measurements; | 18 weeks after baseline
  Body mass index reported as kg/m^2
Ultrasonographic examination; | baseline
  Liver ultrasonography according with criteria by Hamaguchi
Ultrasonographic examination; | 18 weeks after baseline
  Liver ultrasonography according with criteria by Hamaguchi
Glucidic profile | baseline
  fasting glucose reported as mg/dl
Glucidic profile | 18 weeks after baseline
  fasting glucose reported as mg/dl
Insulinemia | baseline
  insulin reported as µU/mL
Insulinemia | 18 weeks after baseline
  insulin reported as µU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Ginanni Corradini, MD, PhD, Principal Investigator — Department Translational and Precision Medicine, Sapienza University of Rome
Locations (1):
- Department of Translational and Precision Medicine, Sapienza University of Rome, Umberto I Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No